CLINICAL TRIAL: NCT04268498
Title: Phase 2, Open-Label Randomized Study of Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone vs Carfilzomib, Lenalidomide, and Dexamethasone in Patients With Newly Diagnosed Multiple Myeloma
Brief Title: A Study of Daratumumab, Carfilzomib, Lenalidomide, and Dexamethasone in Patients With Newly-Diagnosed Multiple Myeloma
Acronym: ADVANCE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: Amgen (Industry); Janssen Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20201316; 2019-001645-41 (EudraCT Number); 19-339 (Other: Memorial Sloan Kettering)
Record Dates: First submitted 2020-02-11; First posted 2020-02-13 (Actual); Last update posted 2025-05-29 (Actual); Status verified 2025-05

CONDITIONS: Multiple Myeloma
Keywords: Daratumumab; Carfilzomib; Lenalidomide
MeSH Terms: conditions — Multiple Myeloma | interventions — Bortezomib; Dexamethasone; Lenalidomide; Acetaminophen; Diphenhydramine; montelukast; carfilzomib; daratumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Arm A - Bortezomib, Lenalidomide and Dexamethasone (VRD) (Experimental): Participants in this group will receive Bortezomib, Lenalidomide and Dexamethasone on a 21 day treatment cycle. Participants achieving a PR or better at the end of 4 cycles will continue to receive a total of 8 cycles of combination therapy. Participants with less than PR after completing 4 cycles will go off study therapy. After 8 cycles of therapy, participants who are MRD positive will have the option to receive an ASCT if stem cells were able to be extracted, before initiating maintenance therapy with Lenalidomide for up to 2 years, and patients who are MRD negative will go directly on to receive maintenance therapy with Lenalidomide for up to 2 years.
  Interventions: Drug: Bortezomib; Drug: Dexamethasone; Drug: Lenalidomide; Biological: Autologous Stem Cell Transplant (ASCT)
- Arm B - Carfilzomib, Lenalidomide and Dexamethasone (KRD) (Experimental): Participants in this group will receive Carfilzomib, Lenalidomide and Dexamethasone on a 28 day cycle. Participants achieving a PR or better at the end of 4 cycles will continue to receive a total of 8 cycles of combination therapy. Participants with less than PR after completing 4 cycles will go off study therapy. After 8 cycles of therapy, participants who are MRD positive will have the option to receive an ASCT if stem cells were able to be extracted, before initiating maintenance therapy with Lenalidomide for up to 2 years, and patients who are MRD negative will go directly on to receive maintenance therapy with Lenalidomide for up to 2 years.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide; Drug: Carfilzomib; Biological: Autologous Stem Cell Transplant (ASCT)
- Arm C- Carfilzomib, Lenalidomide and Dexamethasone with Daratumumab (DKrd) (Experimental): Participants in this group will receive Carfilzomib, Lenalidomide, Dexamethasone with Daratumumab, Acetaminophen, Diphenhydramine and Montelukast on a 28 day cycle. Participants achieving a PR or better at the end of 4 cycles will continue to receive a total of 8 cycles of combination therapy. Participants with less than PR after completing 4 cycles will go off study therapy. After 8 cycles of therapy, participants who are MRD positive will have the option to receive an ASCT if stem cells were able to be extracted, before initiating maintenance therapy with Lenalidomide for up to 2 years, and patients who are MRD negative will go directly on to receive maintenance therapy with Lenalidomide for up to 2 years.
  Interventions: Drug: Dexamethasone; Drug: Lenalidomide; Drug: Acetaminophen; Drug: Diphenhydramine; Drug: Montelukast; Drug: Carfilzomib; Drug: Daratumumab; Biological: Autologous Stem Cell Transplant (ASCT)

INTERVENTIONS:
Drug: Bortezomib — 1.3 mg/m2 administered Subcutaneous (SC) or intravenous (IV) on days 1, 4, 8 and 11 of a 21 day treatment cycle for participants randomized to Arm A.
  Arms: Arm A - Bortezomib, Lenalidomide and Dexamethasone (VRD)
Drug: Dexamethasone — 20 mg or 40 mg per dose administered by mouth (PO) or IV.
  Participants randomized in Arm A:
  20 mg/dose on days 1, 4, 8 and 11 on a 21 day treatment cycle;
  Participants randomized in Arm B:
  Cycles 1 through 8 - 40mg/dose on days 1, 8 and 15 on a 28-day cycle
  Participants randomized in Arm C:
  Cycle 1-2 - 40 mg/dose on days 1, 8, 15 and 22 on a 28-day cycle; Cycles 3-8 - 40mg/dose on Days 1, 8, 15 on a 28-day cycle;
Drug: Lenalidomide — 10 or 25 mg/day capsules administered PO.
  Participants randomized in Arm A:
  25 mg/day capsules on Days 1 through 14 of a 21 day cycle.;
  Participants randomized in Arm B:
  Cycles 1 through 8 - 25 mg/day capsules on Days 1 through 21 of a 28 day cycle;
  Participants randomized in Arm C:
  Cycles 1 - 25 mg/day capsules on Days 2 through 21 of a 28 day cycle; Cycles 2 through 8 - 25 mg/day capsules on Days 1 through 21 of a 28 day cycle;
  Maintenance Therapy:
  10 mg capsules on Days 1 through 21 on a 28 days cycle.
  Other Names: Revlimid
Drug: Acetaminophen — 650 mg administered PO.
  Participants randomized to Arm C:
  Cycles 1 through 8 - 650 mg administered on Days 1, 8 and 15.
  Arms: Arm C- Carfilzomib, Lenalidomide and Dexamethasone with Daratumumab (DKrd)
Drug: Diphenhydramine — 25 mg administered via IV
  Participants randomized to Arm C:
  Cycles 1 through 8 - 25 mg administered on Days 1, 8 and 15.
  Arms: Arm C- Carfilzomib, Lenalidomide and Dexamethasone with Daratumumab (DKrd)
Drug: Montelukast — 10 mg administered PO to participants randomized to Arm C prior to the first 4 doses of Daratumumab.
  Arms: Arm C- Carfilzomib, Lenalidomide and Dexamethasone with Daratumumab (DKrd)
Drug: Carfilzomib — 20 mg or 56 mg/m2 per dose administered via IV.
  Participants randomized to Arm B:
  Cycle 1 - 20 mg/m2 per dose on Day 1 and 56 mg/m2 per dose on days 8 and 15 of a 28 day cycle; Cycles 2 through 8 - 56 mg/m2 per dose on days 1, 8 and 15 of a 28 day cycle;
  Participants randomized to Arm C:
  Cycle 1 - 20 mg/m2 per dose on Day 2 and 56 mg/m2 per dose on days 8 and 15 of a 28 day cycle; Cycles 2 through 8 - 56 mg/m2 per dose on days 1, 8 and 15 of a 28 day cycle
  Arms: Arm B - Carfilzomib, Lenalidomide and Dexamethasone (KRD); Arm C- Carfilzomib, Lenalidomide and Dexamethasone with Daratumumab (DKrd)
Drug: Daratumumab — 16 mg/kg administered via IV or 1800 mg SC, per treating physician discretion.
  Participants randomized to Arm C:
  Cycles 1 though 2 - 16 mg/kg IV or 1800 mg SC on days 1, 8, 15, and 22 of a 28 day cycle; Cycles 3 through 6- 16 mg/kg IV or 1800 mg SC on days 1 and 15 of a 28 day cycle; Cycles 7 through 8 - 16 mg/kg IV or 1800 mg SC on day 1 of a 28 day cycle
  Arms: Arm C- Carfilzomib, Lenalidomide and Dexamethasone with Daratumumab (DKrd)
Biological: Autologous Stem Cell Transplant (ASCT) — Participants who are MRD positive at the conclusion of 8 cycles of study treatment, and were able to have their stem cells that were extracted, will receive ASCT from participants' bone marrow samples.

SUMMARY:
This study is being done to find out whether carfilzomib, lenalidomide, and dexamethasone (KRD) or KRD and Daratumumab (KRD+DARA) might be safer and more effective ways of controlling multiple myeloma than the standard of care treatment, which is lenalidomide, bortezomib, and dexamethasone (VRD).

DETAILED DESCRIPTION:
Per protocol amendment version 4.0 (May 23, 2022), Arm A will be closed and no additional participants will be enrolled in this arm.

ELIGIBILITY:
Inclusion Criteria:

1. Newly diagnosed patients with histologically confirmed Multiple Myeloma (MM) based on the IMWG diagnostic criteria and measurable disease within the past 4 weeks (or past 8 weeks if patient received pre-study MM therapy) based on one of the following:

   * Serum monoclonal protein ≥ 1.0 g/dL
   * Urine monoclonal protein ≥ 200 mg/24 hour
   * Involved serum immunoglobulin free light chain ≥ 10 mg/dL and abnormal kappa/lambda ratio.
2. Evidence of underlying end organ damage and/or myeloma defining event attributed to underlying plasma cell proliferative disorder meeting at least one of the following (Note: Myeloma defining event does not need to be based on repeat testing done at screening, if previous pathology, radiology, etc., confirm diagnosis of myeloma per IMWG)

   * Hypercalcemia: serum calcium >0.25 mmol/L (> 1 mg/dL) above upper limit of normal or ≥ 2.75 mmol/L (11 mg/dL)
   * Anemia: hemoglobin value <10 g/dL or > 2 g/dL below lower limit of normal
   * Bone disease: ≥ 1 lytic lesions on skeletal X-ray, CT, or Positron Emission Tomography (PET)-C. For patients with 1 lytic lesion, bone marrow should demonstrate ≥10% clonal plasma cells
   * Clonal bone marrow plasma cell percentage ≥60%
   * Involved/un-involved serum free light chain ratio ≥100 and involved free light chain

     ≥100 mg/L.
   * > 1 focal lesion on magnetic resonance imaging study (lesion must be >5 mm) in size
   * For patients with 1 lytic lesion, bone marrow should demonstrate ≥10% clonal plasma cells
3. Creatinine Clearance (CrCl) ≥ 60 ml/min. CrCl can be measured or estimated using Cockcroft-Gault method, Modification of Diet in Renal Disease (MDRD), or Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) formulae
4. Age ≥ 18 years at the time of signing the informed consent documentation. Age limit of ≤ 75 years.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-2
6. Absolute neutrophil count (ANC) ≥ 1.0 K/microliter (uL), hemoglobin ≥ 8 g/dL, and platelet count ≥ 75 K/uL, unless if cytopenias are deemed to be due disease at discretion of clinical investigator. Transfusions and growth factors are permissible.
7. Adequate hepatic function, with bilirubin < 1.5 x the pper Limit of Normal (ULN), and Aspartate Aminotransferase (AST) and Alanine Aminotransferase (ALT) < 3.0 x ULN.
8. All study participants must be able to tolerate one of the following thromboprophylactic strategies: aspirin, oral facto Xa inhibitors, low molecular weight heparin, warfarin (coumadin), or alternative anti-coagulant.
9. All study participants must be registered into the mandatory electronic REMS (eREMS) program and be willing and able to comply with the requirements of Risk Evaluation Management and Safety (REMS).
10. Females of childbearing potential (FCBP) must have a negative serum or urine pregnancy test within 10 - 14 days and again within 24 hours prior to prescribing lenalidomide for Cycle 1 (prescriptions must be filled within 7 days) and must either commit to continued abstinence from heterosexual intercourse or begin two acceptable methods of birth control, one highly effective method and one additional effective method at the same time, at least 28 days before she starts taking lenalidomide. FCBP must also agree to ongoing pregnancy testing. Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a successful vasectomy.

A female of childbearing potential is a sexually mature female who: 1) has not undergone a hysterectomy or bilateral oophorectomy; or 2) has not been naturally postmenopausal for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).

Exclusion Criteria:

1. Patients receiving >1 cycle of prior treatment or concurrent systemic treatment for multiple myeloma:

   * Treatment of hypercalcemia or spinal cord compression or aggressively progressing myeloma with current or prior corticosteroids is permitted
   * Bone targeting agents are permitted
   * Concurrent or prior treatment with corticosteroids for indications other than multiple myeloma is permitted
   * Prior treatment with radiotherapy is permitted
   * Prior MM treatments, such as Immunomodulating Drugs (IMIDs) or non-MM drugs in clinical trials for smoldering myeloma is permitted with a washout period of 2 weeks from last dose. Smoldering patients previously treated with carfilzomib are excluded.
   * Patients with measurable disease who received up to one cycle of any therapy within 60 days with a washout period of 2 weeks from last dose (on a trial or outside a trial) are eligible (Note: Measurable disease is defined as one or more of the following: Serum monoclonal protein ≥ 1.0 g/dL, Urine monoclonal protein ≥ 200 mg/24 hour and/ or Involved serum immunoglobulin free light chain ≥ 10 mg/dL AND abnormal kappa/lambda ratio)
2. Prior or current exposure to any of the following:

   * To daratumumab or other anti- Cluster of Differentiation (CD) -38 therapies (unless a re-treatment study)
   * Exposure to an investigational drug (including investigational vaccine) or invasive investigational medical device for any indication within 4 weeks or 5 pharmacokinetic half-lives, whichever is longer.
   * Focal radiation therapy within 14 days prior to randomization with the exception of palliative radiotherapy for symptomatic management but not on measurable extramedullary plasmacytoma.
3. Patients with plasma cell leukemia
4. Patients with Polyneuropathy, Organomegaly, Endocrinopathy, Monoclonal protein, Skin changes syndrome (POEMS syndrome)
5. Patients with amyloidosis
6. Patients with known Chronic Obstructive Pulmonary Disorder (COPD) with a forced expiratory volume in 1 second (FEV1) < 50% of predicted normal. Note that FEV1 testing is required for subjects suspected of having COPD, and subjects must be excluded if FEV1 <50% of predicted normal.
7. Moderate or severe persistent asthma within the past 2 years, or uncontrolled asthma of any classification. Note that participants who currently have controlled intermittent asthma or controlled mild persistent asthma are allowed to participate in the study.
8. Pregnant or lactating females. Because there is a potential risk for AEs in nursing infants secondary to treatment of the mother with carfilzomib in combination with lenalidomide, pregnant or lactating females are excluded from study participation. These potential risks may also apply to other agents used in this study.
9. Uncontrolled hypertension (i.e., systolic blood pressure (BP) >160 mmHg, diastolic BP > 100 mmHg)
10. Uncontrolled diabetes (i.e., two independent glucose readings >200 mg/dL)
11. Active hepatitis B or C infection
12. Subject is:

    * Seropositive for human immunodeficiency virus (HIV)
    * Seropositive for hepatitis B (defined by a positive test for hepatitis B surface antigen [HBsAg]). Subjects with resolved infection (i.e., subjects who are HBsAg negative but positive for antibodies to hepatitis B core (HBc) antigen [anti-HBc] and/or antibodies to hepatitis B surface antigen [anti-HBs]) must be screened using real-time polymerase chain reaction (RT-PCR) measurement of hepatitis B virus (HBV) DNA levels. Those who are PCR positive will be excluded. EXCEPTION: Subjects with serologic findings suggestive of HBV vaccination (anti-HBs positivity as the only serologic marker) AND a known history of prior HBV vaccination do not need to be tested for HBV DNA by PCR.
    * Seropositive for hepatitis C (except in the setting of a sustained virologic response (SVR), defined as aviremia at least 12 weeks after completion of antiviral therapy).
    * Patients with active Coronavirus Disease of 2019 (COVID-19) infection are not to be enrolled until 10 days have passed from the initial positive test, and the patient is symptom-free. COVID-19 vaccinations following national guidelines (i.e., CDC) are encouraged; however, the series should be completed prior to the first day of study treatment. If this is not possible, every effort should be made to administer vaccines at a time when patient is not scheduled to receive study treatment (e.g., "off-weeks").
13. Clinically significant cardiac disease, including:

    * Myocardial infarction within 6 months before randomization, or unstable or uncontrolled disease/condition related to or affection cardiac function (e.g., unstable angina, congestive heart failure, New York Heart Association (NYHA) Class III-IV) or a left ventricular ejection fraction of <40%.
    * Uncontrolled cardiac arrhythmia
    * Intolerance to hydration due to pre-existing pulmonary or cardiac impairment.
14. Pulmonary hypertension
15. Has refractory gastrointestinal (GI) disease with refractory nausea/vomiting, inflammatory bowel disease, or bowel resection that would prevent absorption of oral agents
16. Uncontrolled intercurrent illness including but not limited to active infection or psychiatric illness/social situations that would compromise compliance with study requirements
17. Significant neuropathy ≥ Grade 3 or Grade 2 neuropathy with pain at baseline
18. Contraindication to any concomitant medication, including antivirals or anticoagulation
19. Major surgery within 3 weeks prior to first dose

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Actual)
Dates: Start 2020-02-11 (Actual); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Rate of Minimal Residual Disease (MRD) Negativity | Up to 32 weeks
  MRD will be assessed by the MRD scale ranging from 10 (increased disease detection) to -5 (less to no disease detection) after 8 cycles of therapy.

SECONDARY OUTCOMES:
Overall Survival | Up to 16 weeks
  Overall survival is defined as the time from date of randomization to death from any cause
Progression Free Survival (PFS) | Up to 16 weeks
  PFS is defined as time from date of randomization to time of progression or death, whichever occurs first.
Event Free Survival (EFS) | Up to 16 weeks
  EFS is defined as time from date of randomization to the time of 1) achieving a PR or less with the first four cycles of therapy, 2) transplant, 3) progression, or 4) death, whichever occurs first.
Rate of Response | Up to 3 years
  Rate of Response will be reported as the percentage of participants achieving a response of: a) Partial Response (PR) or better, b) Very Good Partial Response (VGPR) or better and c) Complete Response (CR) and Stringent Complete Response (sCR). Responses will be evaluated from participant serum, urine and bone marrow samples.
Rate of MRD Negativity as best response | Up to 3 years
  MRD will be evaluated from bone marrow samples.
Incidence of treatment related toxicity | Up to 9 months
  Toxicity will be evaluated by treating physician using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) version 5.0.
Minimal Residual Disease (MRD) Negativity | Up to 3 years
  MRD Negativity using bone marrow and blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Carl Landgren, MD, Principal Investigator — University of Miami
Locations (7):
- United States (7):
  - University of Miami, Miami, Florida
  - Moffitt Cancer Center, Tampa, Florida
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Stony Brook University, Stony Brook, New York
  - MD Anderson Cancer Center, Houston, Texas
  - Huntsman Cancer Institue, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No